CLINICAL TRIAL: NCT01685112
Title: Comparison of ECMO Use and Conventional Treatment in Adults With Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201207079RIC
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Septic Shock
Keywords: adults; ECMO
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conventional Group: Patients who developed refractory shock, but didn't received ECMO as salvage treatment
- ECMO group: Patient who have septic shock, and progreseed to have ECMO as salvage therapy

SUMMARY:
Although few cases reported successful treatment of septic shock using extracorporeal membrane oxygenation (ECMO) in adults, no studies compared ECMO to conventional treatment (without ECMO) as treatment for adults with septic shock. Since it is difficult to conduct a randomized study to allocate patients in such critical condition, we aimed to conduct a retrospective observational study using propensity score matched analysis to compare the survival of adults with septic shock treated by ECMO or conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* age >20
* admitted at ICU
* septic shock

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patient who admitted to ICU and had severe sepsis and progressed to septic shock
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | 30 days
  inhospital mortality as primary outcome, mean length of hospital stay around 30 days

CONTACTS AND LOCATIONS:
Overall Officials: YuChung Chuang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan